CLINICAL TRIAL: NCT03872440
Title: ALCMI-012 A Prospective Biospecimen Collection Study From Patients With EGFR Mutant Tumors
Brief Title: PDX Models From EGFR Mutant Tumors
Status: Withdrawn | Type: Observational
Why Stopped: Did not meet the expected enrollment rate.
Sponsor: Addario Lung Cancer Medical Institute (Other)
Responsible Party: Sponsor
Other Study IDs: ALCMI-012
Record Dates: First submitted 2019-01-28; First posted 2019-03-13 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: EGFR mutant cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The purpose of this study is the successful generation of at least ten (10), EGFR mutant PDX models with full characterization including whole exome sequencing (WES) and RNA sequencing. The models will be generated from three major cohorts:
  A.) EGFR T790M patients who have progressed on osimertinib or other third generation (mutant selective) EGFR TKI therapy (n=20) and
  B.) EGFR exon 19 del or L858R patients who have progressed on first line osimertinib (n=20) and
  C.) patients with Exon 20 insertion mutations (n=10; regardless of drug therapy). Includes EGFR Exon 20 and up to two HER2 Exon20 patients.
  The estimates take into consideration an overall take rate of 20%. Models can be used as a resource for clinical and translational research to understand mechanisms of resistance and develop new therapies. For cohort B there is no requirement for a specific number of patients with either EGFR exon 19 deletion or L858R mutations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- EGFR T790M patients: EGFR T790M patients who have progressed on osimertinib or other third generation (mutant selective) EGFR TKI therapy
- EGFR exon 19 del or L858R patients: EGFR exon 19 del or L858R patients who have progressed on first line osimertinib
- Exon 20 insertion mutations patients: Patients with Exon 20 insertion mutations (n=10; regardless of drug therapy). Includes EGFR Exon 20 and up to two HER2 Exon20 patients

SUMMARY:
A biospecimen collection study from individuals with EGFR mutant cancers resistant to EGFR TKIs or those harboring an Exon 20 insertion mutation.

DETAILED DESCRIPTION:
EGFR mutations are detected in approximately 15% of all patients diagnosed with lung cancer. There are several types of EGFR mutations including both the common L858R and exon 19 deletions (accounting for 85%) or the rare exon 20 insertion (accounting for 5-8%) EGFR mutations.

Different types of therapies are being used for these two groups of EGFR mutations. Osimertinib is an EGFR inhibitor approved for patients newly diagnosed with EGFR exon 19 or L858R mutations and for patients who have been treated with a prior EGFR inhibitor but have developed EGFR T790M as a resistance mechanism. In contrast, there are no approved EGFR inhibitors for patients with EGFR or HER2 exon 20 insertion mutations although several therapies are under evaluation in clinical trials.

The Addario Lung Cancer Medical Institute (ALCMI) would like to focus on studying the cancers of patients previously treated with osimertinib or those with EGFR or HER2 exon 20 insertion mutations. The goal is to better understand how these tumors respond to drugs, and what happens when tumors stop responding to drugs. By studying these cancers ALCMI hopes to accelerate the development of new therapeutic approaches for patients with EGFR mutant lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* a. Male or female greater than 18 years of age at the time of consent or the age of majority in their residing state.

  b. Confirmed diagnosis of EGFR mutant NSCLC.
  1. EGFR T790M patients who have progressed on osimertinib or other third generation (mutant selective) EGFR TKI therapy or
  2. Patients must have an EGFR exon 19 deletion or L858R and progressed on first line osimertinib or
  3. Patients with an exon EGFR or HER2 20 insertion mutation.

  c. A clinically-indicated procedure (required by the patient's treating physician) scheduled no more than 30 calendar days from date of consent.

  d. A minimum of 21 calendar days between the last dose of systemic therapy and the clinically-indicated procedure is strongly requested but not required*.

  e. A minimum of 48 hours between the last dose of an osimertinib therapy or other targeted therapies and the time of the clinically-indicated procedure is strongly requested but not required*.

  f. Willingness to undergo all study collection procedures and follow up. g. Provision of written informed consent by the patient. h. Able to communicate (read, write and speak) in English. i. Clinically-indicated procedure to be performed within the US (including Alaska, Hawaii and Puerto Rico), Canada, England, or Israel.

  *A treatment washout period is considered best practice for building a PDX from a tumor specimen. However, if this is not medically possible, material may still be accepted to attempt to build a PDX. This may have a significant impact on take rate therefore accepting tumor specimens with no washout period can impact the overall expected take rate of the program.

Exclusion Criteria:

* a. Less than 18 years of age or age of majority for their residing state, at time of consent.

  b. No confirmed diagnosis of EGFR exon 19 deletion, L858R or EGFR or HER2 exon 20 mutation. Patients whose tumors harbor EGFR mutations other than an exon 19 deletion, L858R or exon 20 EGFR insertion or HER2 exon 20 insertions are not eligible.

  c. A biopsy or surgical procedure not scheduled for clinical/diagnostic purposes.

  d. Pleural effusion specimens collected outside of the US. e. A clinically-indicated procedure scheduled more than 30 calendar days from the date of consent.

  f. Unwilling to undergo all study collection procedures and follow up. g. Unable or unwilling to provide consent. h. Unable to communicate in English. j. Clinically-indicated procedure not scheduled within the US, Canada, England, or Israel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of fifty (50) implantations from approximately fifty (50) subjects, meeting all of the inclusion and none of the exclusion criteria to establish a minimum of ten (10) PDX models.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
The primary objective is to develop a unique cohort of PDX models from EGFR mutant cancers as a resource to the research community. | 48 months
  Successful generation of at least fifty (50) PDX models with full characterization including whole exome sequencing (WES) and RNA sequencing. These PDX models will be used to inform the study of EGFR-driven cancers at large.

CONTACTS AND LOCATIONS:
Locations (1):
- Addario Lung Cancer Medical Institute, San Carlos, California, United States

IPD SHARING:
Plan to Share IPD: No